CLINICAL TRIAL: NCT00032500
Title: Evaluation of Echinacea in a Human Rhinovirus Challenge
Brief Title: Evaluation of Echinacea for the Common Cold
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01AT001146-01 (NIH)
Record Dates: First submitted 2002-03-22; First posted 2002-03-25 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Common Cold
Keywords: common cold; Echinacea
MeSH Terms: conditions — Common Cold | interventions — Echinacea extract

INTERVENTIONS:
Drug: Echinacea

SUMMARY:
The purpose of this study is to determine whether three Echinacea preparations with different chemical compositions are effective for prevention or treatment of the common cold.

DETAILED DESCRIPTION:
Echinacea is a widely used herbal remedy for the common cold. Previous clinical trials designed to assess the efficacy of Echinacea for prevention or treatment of the common cold have produced inconsistent results. A variety of different Echinacea products have been used in these clinical trials. Recent studies indicate that different Echinacea preparations have dramatically different phytochemical profiles. The available clinical trial data provide no information about the potential role of the different constituents of Echinacea in common cold prevention or treatment. Our hypothesis is that the variation in reported clinical effectiveness may be due to differences in the phytochemical profile of the Echinacea preparations used. This study will address the following specific aims: 1) Evaluate the effectiveness of chemically defined extracts of E. angustifolia root which contain alkamides, echinacoside or polysaccharidelglycoprotein for common cold prevention or treatment; 2) Assess the correlation between specific Echinacea metabolites in serum and nasal secretions and efficacy for prevention and treatment of colds; and 3) Determine the effect of different Echinacea preparations on the host response to rhinovirus infection.

Age Groups: Child, Adult, Older Adult
Dates: Start 2001-09; Study Completion 2004-05

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B. Turner, MD, Principal Investigator — University of Virginia School of Medicine; J. David Gangemi, PhD — Clemson University; Rudolf Bauer, PhD — Karl-Franzens-Universitaet Graz
Locations (1):
- University of Virginia, Charlottesville, Charlottesville, Virginia, United States

REFERENCES:
- [Result] Turner RB, Bauer R, Woelkart K, Hulsey TC, Gangemi JD. An evaluation of Echinacea angustifolia in experimental rhinovirus infections. N Engl J Med. 2005 Jul 28;353(4):341-8. doi: 10.1056/NEJMoa044441. PMID 16049208